CLINICAL TRIAL: NCT05025150
Title: Point-of-Care Ultrasound for Pediatric Thoracic Trauma: A Multi-Institutional Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, HIU FUNG SAMUEL LAM, Attending physician, Sutter Health
Other Study IDs: 2019.091EXP
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Trauma Chest; Pediatric ALL
Keywords: Ultrasonography
MeSH Terms: conditions — Thoracic Injuries; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the proposed study is to investigate the diagnostic accuracy of ED POCUS in pediatric traumatic thoracic injuries including traumatic pneumothorax, hemothorax, lung contusion, rib fractures, and pulmonary edema (from submersion injury). This will be a prospective, multicenter, observational study of children 0-21 years of age presenting to the participating pediatric emergency departments for suspected traumatic thoracic injury. Results of POCUS will be compared to that of chest X-ray, final clinical diagnosis, computed tomography (CT) or magnetic resonance imaging (MRI). Study hypotheses are that POCUS is highly accurate (90-95%) when compared to chest X-ray, and moderately accurate (~80%) when compared to CT or MRI in diagnosing these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be children 0 to 21 years of age presenting to the participating PEDs meeting trauma activation criteria and with suspected thoracic injury.

Exclusion Criteria:

* Congenital or acquired cardiopulmonary or osteogenic conditions rendering POCUS ineffective, foreign body/ barrier to lung ultrasound of which removal is contraindicated, subjects under law-enforcement custody, and subjects deemed unsuitable by treating clinicians.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Suspected penetration injury to neck, chest or abdomen
  * Falls >10 feet or more than 3 times of the child's height
  * Suspected spinal cord injury with neurological deficits
  * Pedestrian or cyclist hit or run over by car at >20mph
  * Motor vehicle collision (MVC) at high speed >50mph or with ejection of occupant
  * MVC with death of another occupant or prolonged extrication time or significant intrusion to passenger compartment.
  * Crash or flip of motorized vehicle with separation of rider from vehicle
  * High voltage electrical injury (>220V)
  * Hanging
  * Submersion injury
  * Trauma mechanism with cardiac arrest or hypotension adjusted for age
  * Explosion injury
  * Treating physician discretion on patients otherwise not meeting any of the above criteria
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of POCUS as compared to chest X-ray in detecting injuries | 7-10 days

SECONDARY OUTCOMES:
Compare the accuracy of POCUS to cross sectional imaging (CT or MRI). | 7-10 days
Compare the accuracy of POCUS to chest X-ray or final clinical diagnosis (if no other imaging is performed). | 7-10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sutter Medical Center Sacramento, Sacramento, California, United States